CLINICAL TRIAL: NCT03461939
Title: Electronic Patient Self-Reported Outcomes to Improve Cancer Management and Patient Experiences (ePRIME): Collection of Patient-reported Adverse Events in Early Phase Clinical Trials in Yorkshire
Brief Title: ePRIME: Patient-Reported AEs in Early Phase Trials
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: Yorkshire Cancer Research (Other); The Leeds Teaching Hospitals NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Galina Velikova, Professor of Psycho-social and Medical Oncology/Consultant in Medical Oncology, University of Leeds
Other Study IDs: L392 (EPT)
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cancer
Keywords: ePRIME; PRO; PROM; Adverse event; QTool; Early phase; CTCAE
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ePRIME: Participants in the study will receive training in using the ePRIME system to report their symptoms and side effects on a weekly basis from home via the internet for 12 weeks while receiving early phase trial treatment. Patients will be sent email/text reminders to enter their symptoms on the system once a week. Patients will be reminded that the data they enter via the online system will not be reviewed promptly by their hospital team and therefore they should continue to contact their treatment team via the contact numbers they have been given.
  As part of the research project, we will monitor the number of notifications for severe AE generated by the system to address concerns from the interviews conducted in the first phase of this research project that ePROs will lead to increased workload for clinicians.
  Interventions: Other: ePRIME symptom monitoring tool

INTERVENTIONS:
Other: ePRIME symptom monitoring tool — ePRIME is an online system for patients to self-report symptoms and AE during cancer treatment. ePRIME allows AE reporting from home or hospital and enables patient reported data to be integrated into existing EPR to allow for the reports to be used in routine care. In addition the system is capable of generating notifications for severe AE to the relevant clinical team and providing patient advice on managing mild and moderate AE.

SUMMARY:
New treatments are continually being developed to help patients living with advanced cancer, which require extensive clinical trials before authorisation for standard clinical use. Reporting of adverse events (AE) in this setting is essential to ensure treatment safety and tolerability. The current system for reporting AEs, the Common Toxicity Criteria and Adverse Events (CTCAE) relies on the clinician's interpretation of patient symptoms, but a substantial body of evidence suggests clinicians miss/underestimate AEs experienced by patients. The aim of the overall project is to explore the implementation of an electronic patient-reported outcomes (ePRO) system to gather adverse events data in early phase clinical trials (EPCT) patients. In Phase 1 of this study, through semi-structured interviews, we explored patient, healthcare, and clinical trial staffs' views about collecting electronic patient-reported outcomes in this setting. This work informed the direction of the current pilot. This proof-of-principle feasibility study will explore the feasibility and satisfaction with using an electronic system to remotely self-report AEs whilst on EPCT. The key objectives are to:

1. Evaluate the feasibility of using a secure online method (ePRIME system) to collect PRO-AEs in EPCT patients.
2. Explore patient satisfaction with the use of the ePRIME system to collect PRO AEs in EPCT patients.
3. Monitor the number of notifications for severe AEs generated by the system to address concerns from the interviews that ePROs will lead to increased workload.

To this end, a prospective longitudinal pilot will be conducted of the ePRIME system in early phase clinical trial patients in Leeds and Sheffield. A convenience sample of patients enrolled in Phase I or Phase II trials will be recruited. Patients in general oncology and haematology clinics will be included if diagnosed with metastatic or progressive disease and are presently receiving novel agents in an academic early phase clinical trial, such as chemotherapy, targeted agents, or chemo-radiotherapy. Patients will be included in this pilot whether the trial is a test of a novel drug, drug combination, or dose escalation. The study will aim to identify, approach, and consent all eligible patients over a minimum of a 12 month period. If they are over 18, able to give informed consent, have access to internet via any device, and able to read and understand English. Patients will be approached and consented within 1 month of having been entered in the clinical trial. Patients will not be eligible if they will be on the clinical trial for less than 3 months. Each patient will complete a patient-reported AE checklist at baseline (i.e. time of consent) and then weekly for 12 weeks. At the end of the 12 weeks an end-of-study interview will be conducted to explore patient satisfaction with the system. It is envisaged that this project will provide initial information on the feasibility and acceptability of a novel electronic system to facilitate the collection of patient-reported AEs in early phase trials.

ELIGIBILITY:
Inclusion Criteria

* Cancer patients enrolled in an academic Phase I or Phase II EPCT;
* Patients receiving novel anticancer agents, including but not limited to novel agents, such as chemotherapy, targeted agents, or chemo-radiotherapy, chemo-immunotherapy ;
* Within 1 month of having started treatment on an early phase clinical trial;
* Able and willing to give informed consent;
* Able to read and understand English;
* Access to internet via a computer, laptop, tablet or mobile phone;
* Aged ≥ 18.

Exclusion Criteria

* Patients involved in an EPCT involving surgery or radiotherapy alone;
* Patients involved in commercial EPCTs
* Patients who will be on an early phase clinical trial for less than 3 months;
* Evidence of overt psychopathology or serious cognitive dysfunction which would impede study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled and receiving treatment on a early phase clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of using a secure, online system to record, monitor, and help patients report AEs. | 2018-2020
  Feasibility of using a secure, online system to record, monitor, and help patients report AEs. It will be measured through:
  * the number of participants consenting versus declining;
  * compliance with the ePRIME trial through the number of missed completions, out of the 12 weeks (minimum) prompted by the research team;
  * number and timing of participant withdrawals and reasons;
  * number of completions in addition to the weekly prompts;
  * number of completions that generate notifications to the early phase clinical trials ePRIME email address.

SECONDARY OUTCOMES:
Participant satisfaction with using the system | 2018-2020
  We will explore participant satisfaction with the use of the system. Through an end-of-study interview with patients and healthcare professionals we will explore the perceived burden, barriers, and opportunities and benefits of using the novel system. In addition to this, we will also explore system usability parameters such as time of log-on and log-off, time taken to complete the measures, time outs, and time spent on each page/section.

CONTACTS AND LOCATIONS:
Overall Officials: Galina Velikova, Principal Investigator — University of Leeds
Locations (2):
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shearsmith L, Danson S, Gelcich S, Gibson A, Gordon K, Collinson F, Croft J, Griffiths E, Rogers Z, Carter R, Brown J, Velikova G, Kennedy F. Electronic patient-reported adverse event monitoring in academic early-phase clinical trials: A feasibility study. Clin Trials. 2025 Oct 27:17407745251378668. doi: 10.1177/17407745251378668. Online ahead of print. PMID 41140127
- See also: Research group website/webpage relating to the study — http://www.pogweb.org/index.php/eprime/